CLINICAL TRIAL: NCT06220799
Title: Impact of the Craniovertebral Angle on the Cervicogenic Dizziness and the Risk of Falling in Patients With Cervical Radiculopathy
Brief Title: Impact of Craniovertebral Angle on Dizziness and Risk of Falling in Cervical Radiculopathy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Abdelrahman Elsayed Hassan Aboud, Teaching assistant of physical therapy for neuromuscular disorders and its surgeries, Cairo University
Other Study IDs: P.T.REC/012/004743
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Study group (GI): The Study group (GI) will include twenty five patients with chronic cervical radiculopathy with forward head posture (FHP) (CVA=less than 49° ).
- The Control group (GII): The Control group (GII) will include twenty five patients with chronic cervical radiculopathy without forward head posture (FHP)( CVA = more than 49).

SUMMARY:
-The goal of this observational study is to learn about the impact of the changes in cranio-vertebral angle on the cervicogenic dizziness and the risk of falling in the patients with cervical radiculopathy .The main question it aims to answer is: Is there an impact of the changes in cranio-vertebral angle on the cervicogenic dizziness and the risk of falling in the patients with cervical radiculopathy ? The participants will be undergone measuring the cranio-vertebral angle ,assessment of cervical proprioception and other tasks and questions through 3scales .

Researchers will compare between study group and control group to see if there isimpact of the changes in cranio-vertebral angle on the cervicogenic dizziness and the risk of falling in the patients with cervical radiculopathy .

ELIGIBILITY:
Inclusion Criteria:

* The Patients will include if they have the following:

  1. Fifty patients with chronic cervical radiculopathy(degenerative type) from both sex will participate in the study (twenty five with forward head posture (FHP) , and twenty five without forward head posture (FHP) ).
  2. The duration of the disease (cervical radiculopathy)is more than 6 months.
  3. The age ranged from 35 to 50 years old.
  4. Mild to moderate neck pain on visual analogue scale .
  5. Pain and dizziness lasting for 3-6 months.
  6. subjective dizziness experienced in conjunction with cervical pain, movement, stiffness, or particular postures.

     Exclusion Criteria:
* The Patients will exclude if they exhibit any of the following:

  1. Cervical myelopathy.
  2. Cervical myelo-radiculopathy.
  3. Acute cervical radiculopathy.
  4. Diabetic neuropathy.
  5. Previous cervical surgery.
  6. Cervical trauma.
  7. Deformities in the cervical spine .
  8. Rheumatoid arthritis.
  9. Any tumours and infection involving the cervical spine .
  10. Patients with a history of neuromuscular disorders.
  11. precise diagnosis of either central dizziness (due to cerebrovascular disorders related to the vertebrobasilar circulation, migraine, multiple sclerosis, tumours of the posterior fossa, neurodegenerative disorders, some drugs, and psychiatric disorders) or peripheral dizziness( due to a problem in the part of the inner ear that controls balance. These areas are called the vestibular labyrinth, or semicircular canals. The problem may also involve the vestibular nerve. This is the nerve between the inner ear and the brain stem).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fifty patients with chronic cervical radiculopathy(degenerative type) from both sex will be enrolled in this study. Patients will be assigned into two groups (study and control groups) . The Study group (GI) will include twenty five patients with chronic cervical radiculopathy with forward head posture (FHP) (CVA=less than 49° ). Control group (GII) will include twenty five patients with chronic cervical radiculopathy without forward head posture (FHP)( CVA =more than 49°). Patients in group I were diagnosed as patients with chronic cervical radiculopathy with forward head posture (FHP) based on careful clinical evaluation by the neurologist . The patients will be recruited from the faculty of Physical Therapy, Cairo University, and private clinic in cairo .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-01-29 (Estimated); Study Completion 2024-01-29 (Estimated)

PRIMARY OUTCOMES:
Craniovertebral angle (CVA) | 20 minutes
  Taking photos from lateral view then craniovertebral angle measured by Kinovea software program.
Cervical joint position error . | 40 minutes
  Cervical joint position error via the CROM device,through the neutral head repositioning test (NHR) and the target head repositioning test (THR).
Cervicogenic dizziness. | 10 minutes
  Cervicogenic dizziness via score of Dizziness Handicap Inventory Questionnaire(DHI).
The risk of falling. | 20 minutes
  The risk of falling assessed by Berg Balance Scale(BBS) .
The fear of falling. | 10 minutes
  The fear of falling assessed by Fall Efficacy Scale-International(FES-I).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Labs at Cairo University, Dokki, Giza Governorate, Egypt